CLINICAL TRIAL: NCT05722964
Title: Efficacy and Safety of Intravenous Infusion of SHR-1906 in Patients With Idiopathic Pulmonary Fibrosis: a Multicenter, Randomized, Double-blind, Parallel Placebo-controlled Phase II Trial
Brief Title: Study on Intravenous Injection of SHR-1906 in the Treatment of Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1906-201
Record Dates: First submitted 2023-01-11; First posted 2023-02-10 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Comparison of SHR-1906 injection and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1906，-Dose A (Experimental)
  Interventions: Drug: SHR-1906
- SHR-1906，- Dose B (Experimental)
  Interventions: Drug: SHR-1906
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1906 — Intravenous injection
  Arms: SHR-1906，-Dose A
Drug: SHR-1906 — Intravenous injection
  Arms: SHR-1906，- Dose B
Drug: Placebo — Placebo，Intravenous injection
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of intravenous SHR-1906 in the treatment of idiopathic pulmonary fibrosis. The study is divided into four stages: screening period, baseline period, treatment period and safe follow-up period. It is planned that 108 patients will be randomly assigned to the following three treatment groups for treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 to 80, inclusive, at the time of screening；
2. IPF diagnosed according to ATS/ERS/JRS/ALAT guidelines (2022) (HRCT diagnosis UIP type/possible UIP type (standard HRCT confirmed by central review in recent 3 months) with or without pathological UIP type/possible UIP type (pathology refers to frozen lung biopsy or surgical/thoracoscopic lung biopsy)；
3. 90% ≥ FVCpp ≥ 45% during screening period and the first day;
4. The percent of predicted DLCO value (corrected by Hb value) at screening is ≥ 30% and ≤ 90%;
5. Before the screening period, pirfenidone or nidanib with stable dose ≥ 8 weeks (pirfenidone ≥ 1200 mg/denidanib ≥ 200 mg/d) can continue to maintain treatment with stable dose during the study period; Or at least 4 weeks before the screening period, pirfenidone or nidanib was not used (pirfenidone or nidanib was refused due to intolerance or various factors) ；

Exclusion Criteria:

1. Evidence of any of the following significant obstructive pulmonary disease: (1) The ratio of forced expiratory volume/forced vital capacity (FEV1/FVC) at the first second is < 0.70 (after using bronchodilator) or (2) HRCT shows that emphysema is greater than fibrosis;
2. Interstitial lung diseases (ILD) other than IPF include but are not limited to: any other type of idiopathic interstitial pneumonia; Lung diseases related to contact with fibroblasts or other environmental toxins or drugs; Other types of occupational lung diseases; Granulomatous lung disease; Pulmonary vascular disease; Systemic diseases include vasculitis infectious diseases (i.e. Tuberculosis) and connective tissue diseases If the diagnosis is unclear, serological examination and/or multidisciplinary expert group review should be conducted to confirm IPF or other types of ILD diagnosis;
3. A history of other types of respiratory diseases, including respiratory tract, lung parenchyma, pleural cavity, mediastinum, diaphragm or chest wall diseases or disorders, such as acute respiratory infection, active tuberculosis, etc., which researchers believe will affect the primary endpoint of the study or otherwise affect the participation of subjects in the study;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in FVC% (Percent of Predicted FVC value) to week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Change from Baseline in FVC (L) to Week 4, 8, 12, 16, 20, 24 | Baseline, Week 4, 8, 12, 16, 20, 24
Change from Baseline in FVC% (Percent of Predicted FVC value) to Week 4, 8, 12, 16, 20 | Baseline, Week 4, 8, 12, 16, 20
Change from Baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) to Week 12 and Week 24 | Baseline, Week 12 and Week 24
Change from Baseline in St. George's Respiratory Questionnaire (SGRQ) Scores to Week 12 and Week 24 | Baseline, Week 12 and Week 24]
Number of Praticipants with an Acute Exacerbation of IPF | Start of Treatment to end of study (approximately 28 weeks)
All-cause mortality | Start of Treatment to end of study (approximately 28 weeks)
Adverse events | Start of Treatment to end of study (approximately 28 weeks)
Serum concentration of SHR-1906 | Start of Treatment to end of study (approximately 28 weeks)
Proportion of anti-SHR-1906 antibody (ADA) formed during the study from baseline | Start of Treatment to end of study (approximately 28 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided